CLINICAL TRIAL: NCT04060082
Title: VOICE Of bvFTD [Voices Of Individuals: Challenges and Experiences Of bvFTD]
Brief Title: Voices Of Individuals: Challenges and Experiences Of bvFTD
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 833507
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Frontotemporal Dementia; Frontotemporal Degeneration; Frontotemporal Dementia, Behavioral Variant; FTD
Keywords: FTD; Interview; Genetics; Persons diagnosed; Frontotemporal degeneration; bvFTD; Chromosome 9 open reading frame 72 (C9ORF72); Microtubule-associated protein tau (MAPT); Progranulin (GRN); TAR DNA-binding protein (TARDBP); Valosin-Containing Protein (VCP); Charged multivesicular body protein 2B (CHMP2B)
MeSH Terms: conditions — Frontotemporal Dementia; Pick Disease of the Brain; Frontotemporal Dementia With Motor Neuron Disease; Inclusion Body Myopathy With Early-Onset Paget Disease And Frontotemporal Dementia | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Persons Diagnosed: Individuals with a diagnosis of bvFTD.
  Interventions: Other: Telephone Interview
- Persons At Risk: Individuals with a known genetic risk factor for bvFTD: people with genetic testing that identified a disease-causing change in a gene that is known to cause bvFTD, such as in C9ORF72, MAPT, GRN, VCP, TARDBP, CHMP2B, or another gene that has been identified as causing FTD in the family
  Interventions: Other: Telephone Interview

INTERVENTIONS:
Other: Telephone Interview — Participants will be asked to answer questions about their experiences with FTD.

SUMMARY:
The VOICE Of bvFTD study is a telephone interview research study about life with or at risk for behavioral variant frontotemporal dementia (bvFTD). The study aims to understand how bvFTD impacts individuals' day to day lives, how people think about themselves, and what challenges they face.

DETAILED DESCRIPTION:
The VOICE Of bvFTD study is a study being conducted at the University of Pennsylvania. The study was developed and initiated in collaboration with the Johns Hopkins Bloomberg School of Public Health and the National Human Genome Research Institute. The goal of this study is to learn more about what it is like to live with or at high risk of developing behavioral variant frontotemporal dementia (bvFTD). The study will involve telephone interviews to help learn as much as possible about living with bvFTD. The hope is that this will guide future research, resource development, and clinical practice.

Participants will have at least two phone calls from the study team. During the initial phone call, which will take about 15 to 20 minutes, the participant will be asked some basic questions about demographics and the study details will be reviewed as part of the consent process. During another call the participant will be asked some questions to assess his or her thinking, and will complete the interview which will last about 30 to 60 minutes. There are no physical or medical procedures included in this study. The consent process, screening, interview scheduling, and the interview itself will take place over two or three phone calls, which may occur over several weeks.

A person may be able to take part in this study if they are a person with bvFTD, or if they have been found to have a genetic change that causes bvFTD.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Speak fluent English
* People with bvFTD must have been diagnosed with behavioral variant frontotemporal degeneration (bvFTD)
* People with a known genetic risk factor for bvFTD must have an identified disease-causing change in a gene that is known to cause bvFTD, such as in C9ORF72, MAPT, GRN, VCP, TARDBP, CHMP2B, or another gene that has been identified as causing FTD in the family
* The diagnosis or genetic testing results must have been disclosed to the participant at least two months prior to study enrollment

Exclusion Criteria:

* Inability to complete the informed consent comprehension process
* Under 18 years of age
* Does not speak English
* Received diagnosis or testing result less than two months prior to study enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants for the study will be recruited through the University of Pennsylvania and ClinicalTrials.gov. Previously, participants were also recruited through Johns Hopkins University, through a dementia research study at the National Institutes of Health, through the Penn FTD Center Caregiver Conference, and through through a private Facebook group for individuals with C9orf72 mutations.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Affective and Behavioral Responses | Through study completion: about 1.5-2 hours total over several weeks
  How participants describe and categorize their emotional reactions to receiving a diagnosis of bvFTD or positive genetic testing result, and their experiences living with that knowledge. It will also explore how patients describe their behavior in response to the testing or diagnosis, such as use of coping strategies, challenges faced, and decisions to disclose their status to family and friends.

CONTACTS AND LOCATIONS:
Overall Officials: Jill Owczarzak, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Lori Erby, PhD, ScM, Principal Investigator — National Institutes of Health (NIH)
Locations (3):
- United States (3):
  - Johns Hopkins Medical Institution, Baltimore, Maryland
  - National Institutes of Health (NIH), Bethesda, Maryland
  - University of Pennsylvania (Penn Frontotemporal Degeneration Center), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No